CLINICAL TRIAL: NCT04003220
Title: Idiopathic Chronic Thrombocytopenia of Undetermined Significance : Pathogenesis and Biomarker
Acronym: ICTUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/47
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Thrombocytopenia; Purpura, Thrombocytopenic; Myelodysplastic Syndromes
MeSH Terms: conditions — Thrombocytopenia; Purpura, Thrombocytopenic; Myelodysplastic Syndromes | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the samples for research will be taken in the department where the patient is:
  * Blood sampling: 5 ACD-A tubes (Acid Citrate Dextrose) and 2 EDTA tubes (for 30 ICTUS patients, 20 ITP patients, and 20 patients with MDS)
  * One supplementary tube of bone marrow (for 10 patients with ICTUS, and 10 Healthy controls)
  * 25 Hair bulbs (for 20 ICTUS patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MyeloDysplastic Syndrome: platelets <150 G/l and diagnosis of myelodysplasia according to the WHO classification (abnormal bone marrow features).
  Interventions: Procedure: blood sample
- Idiopathic Chronic Thrombocytopenia of Unknown Significance: Acquired thrombocytopenia lasting>6 months, without feature of dysimmunity (antiplatelet Ab, or anti nuclear Ab, anti ENA Ab, ANCA, anti-CCP Ab, cryoglobulinemia), normal bone marrow examination, absence of other thrombocytopenia in the family. All ICTUS patients included in the study will thus have a bone marrow aspiration.
  Interventions: Procedure: blood sample; Procedure: Bone marrow sample
- Immune Thrombocytopenic Purpura: Diagnosis of Immune Thrombocytopenic Purpura (ITP) is made according to the international ITP consensus (diagnostic criteria of Rodeghiero){Provan, 2010 #18}, knowing that a presumptive diagnosis of ITP is made when the history, physical examination, complete blood count, and examination of the peripheral blood smears do not suggest other etiologies for the thrombocytopenia
  Interventions: Procedure: blood sample
- healthy volunteers undergoing cardiac surgery: patients with normal blood counts undergoing cardiovascular surgery for valve replacement, or healthy bone-marrow donors
  Interventions: Procedure: Bone marrow sample

INTERVENTIONS:
Procedure: blood sample — The extra samples will be taken Blood sampling
  Groups: Idiopathic Chronic Thrombocytopenia of Unknown Significance; Immune Thrombocytopenic Purpura; MyeloDysplastic Syndrome
Procedure: Bone marrow sample — This bone marrow sampling will be performed for 10 patients with ICTUS, and 10 controls
  Groups: Idiopathic Chronic Thrombocytopenia of Unknown Significance; healthy volunteers undergoing cardiac surgery

SUMMARY:
It is a translational research study with mechanistical objectives and including biological samples of patients with thrombocytopenia

DETAILED DESCRIPTION:
This study is a prospective study to collect blood, bone marrow and hair bulb from patients with thrombocytopenia, to better understand the mechanism of idiopathic chronic thrombocytopenia of undetermined significance (ICTUS)

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80
* Nosological criteria for thrombocytopenic patients:
* ICTUS: acquired thrombocytopenia lasting>6 months, without feature of dysimmunity (antiplatelet Ab, or anti nuclear Ab, anti ENA Ab, ANCA, anti-CCP Ab, cryoglobulinemia), normal bone marrow examination, absence of other thrombocytopenia in the family. All ICTUS patients included in the study will thus have a bone marrow aspiration.
* ITP: Diagnosis of ITP is made according to the international ITP consensus (diagnostic criteria of Rodeghiero){Provan, 2010 #18}, knowing that a presumptive diagnosis of ITP is made when the history, physical examination, complete blood count, and examination of the peripheral blood smears do not suggest other etiologies for the thrombocytopenia. There is no "gold standard" test that can reliably establish the diagnosis. We are concerned that this group of patients may include ICTUS patients.
* ITP with immunological features: ITP with detectable anti-platelet antibodies (Ab) and/or autoimmunity (anti nuclear Ab, anti ENA Ab, ANCA, anti-CCP Ab, cryoglobulinemia), and/or previously responsive to immunomodulatory ITP-directed therapies (steroids, intravenous Immunoglobulin, rituximab, splenectomy). We will use these patients as non-ICTUS, ITP positive controls.
* Thrombocytopenic myelodysplasia: platelets <150 G/l and diagnosis of myelodysplasia according to the WHO classification (abnormal bone marrow features).
* Healthy controls: patients with normal blood counts undergoing cardiovascular surgery for valve replacement, or healthy bone-marrow donors.
* Affiliated person or beneficiary of a social security scheme. Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Age under 18 or over 80
* Persons placed under judicial protection,
* Persons participating in another research including a period of exclusion still in course
* Persons in emergency situation,
* Pregnant or nursing women,
* Women of childbearing age who do not benefit from effective contraception (HAS criteria),
* Brain death or deceased persons,
* Person who doesn't speak French, doesn't read it, doesn't write it, and doesn't have a schooling in France.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this project we will study 30 patients with ICTUS, 20 ITP with immunological features, 20 MDS patients and 10 Healthy volunteers (normal bone marrow donors, obtained during a sternotomy performed in the cardiac surgery unit).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-09-07 (Estimated); Study Completion 2023-09-07 (Estimated)

PRIMARY OUTCOMES:
Measure of clonality in patients with ICTUS | Day 1
  identification of mutations in genes known to be involved in clonal expansion

CONTACTS AND LOCATIONS:
Overall Officials: JAMES, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (4):
- France (4):
  - Immunopathologie Clinique - Hôpital Saint Louis - AP HP, Paris
  - Chirurgie cardiaque - Hôpital Haut Lévêque - CHU de Bordeaux, Pessac
  - Service des maladies du sang - Hôpital Haut-Lévêque - avenue de Magellan, Pessac
  - service de médecine interne et maladies infectieuses - Groupe hospitalier Sud, Pessac

IPD SHARING:
Plan to Share IPD: No